CLINICAL TRIAL: NCT05187169
Title: An Open-Label, 2-Way, 2-Period Crossover Study of Orally Administered VS-6766 in Healthy Adult Subjects to Determine the Effect of Food on the Pharmacokinetics of VS-6766
Brief Title: Food Effect of VS-6766 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VS-6766-101
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Food Effect

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, 2-way, 2-period crossover, Food Effect study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Active Comparator): 4.0 mg VS-6766, following an overnight fast of at least 10 hours
  Interventions: Drug: VS-6766
- Treatment B (Active Comparator): 4.0 mg VS-6766, administered 30 minutes after the start of a high-fat/high-calorie meal breakfast
  Interventions: Drug: VS-6766

INTERVENTIONS:
Drug: VS-6766 — Dual RAF/MEK inhibitor

SUMMARY:
An Open-Label, 2-Way, 2-Period Crossover Study of Orally Administered VS-6766 in Healthy Adult Subjects to Determine the Effect of Food on the Pharmacokinetics of VS-6766

DETAILED DESCRIPTION:
This is an open-label, randomized, 2-way, 2-period crossover, Food Effect study.

On Day 1 of each period, subjects will receive a single oral dose of VS-6766 administered in a 2-way crossover fashion either under fasting conditions or following a standardized high-fat/high-calorie meal. PK sampling for VS-6766 will be collected predose and postdose. There will be a washout period between doses.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female (of non-childbearing potential only), 18-55 years of age, inclusive, at the screening visit.
2. Must follow protocol specified contraception guidance.
3. Continuous non-smoker who has not used tobacco/nicotine-containing products for at least 3 months prior to the first dosing based on subject self-reporting.
4. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at the screening visit.
5. Medically healthy with no clinically significant medical history.
6. Able to swallow capsules.
7. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Presence of systemic or severe infection.
2. History or presence of a significant medical condition or disease which is not completely resolved.
3. History or presence of alcohol or drug abuse
4. History or presence of hypersensitivity or reaction to the study drug or related compounds.
5. History of tuberculosis.
6. Presence of any fever within 2 weeks prior to first dosing.
7. Females able to have children.
8. Females who are pregnant or lactating.
9. Presence of HIV.
10. Must be able to refrain from using any drugs, including prescription and non-prescription medications beginning 28 days prior to the first dosing.
11. Lactose Intolerance.
12. Donation of blood or significant blood loss or blood transfusion within 56 days prior to the first dosing.
13. Plasma donation within 7 days prior to the first dosing.
14. Participation in another clinical study within 30 days prior to the first dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Plasma Pharmacokinetics (PK) of a single dose of VS-6766 after a standardized high-fat/high-calorie meal and after fasting: AUC0-t | 30 days
  Area under plasma Concentration (AUC) 0 to t
Plasma Pharmacokinetics (PK) of a single dose of VS-6766 after a standardized high-fat/high-calorie meal and after fasting: AUC0-120 | 30 days
  Area under plasma Concentration (AUC) from 0-120 minutes
Plasma Pharmacokinetics (PK) of a single dose of VS-6766 after a standardized high-fat/high-calorie meal and after fasting: AUC0-inf | 30 days
  Area under plasma Concentration (AUC) from zero to infinity
Plasma Pharmacokinetics (PK) of a single dose of VS-6766 after a standardized high-fat/high-calorie meal and after fasting: AUC%extrap | 30 days
  Area under plasma Concentration (AUC) extrapolated
Plasma Pharmacokinetics (PK) of a single dose of VS-6766 after a standardized high-fat/high-calorie meal and after fasting: Cmax | 30 days
  Cmax for VS-6766 administered with and without food.
Plasma Pharmacokinetics (PK) of a single dose of VS-6766 after a standardized high-fat/high-calorie meal and after fasting: Tlag | 30 days
  absorption lag-time (Tlag)
Plasma Pharmacokinetics (PK) of a single dose of VS-6766 after a standardized high-fat/high-calorie meal and after fasting: Tmax | 30 days
  time of Maximum concentration (Tmax)
Plasma Pharmacokinetics (PK) of a single dose of VS-6766 after a standardized high-fat/high-calorie meal and after fasting: Kel | 30 days
  Elimination rate (Kel)
Plasma Pharmacokinetics (PK) of a single dose of VS-6766 after a standardized high-fat/high-calorie meal and after fasting: T1/2 | 30 days
  concentration Half-life (T1/2)
Plasma Pharmacokinetics (PK) of a single dose of VS-6766 after a standardized high-fat/high-calorie meal and after fasting: CL/F | 30 days
  Oral Clearance (CL/F)
Plasma Pharmacokinetics (PK) of a single dose of VS-6766 after a standardized high-fat/high-calorie meal and after fasting: Vz/F | 30 days
  Apparent Volume of Distribution (Vz/F) for VS-6766 administered with and without food.

SECONDARY OUTCOMES:
To assess the safety and tolerability of a single-dose of VS-6766 administered with or without a standardized high-fat/high-calorie meal in healthy adult subjects. | 30 days
  Treatment emergent adverse events/ treatment emergent serious adverse events - their frequency, duration and severity, lab parameters, vital signs, ECG and ophthalmologic changes

CONTACTS AND LOCATIONS:
Overall Officials: Louis Denis, MD, Study Director — Verastem, Inc.
Locations (1):
- Celerion, Tempe, Arizona, United States